CLINICAL TRIAL: NCT05319873
Title: A Phase 1B Trial Evaluating the Safety of Ribociclib, Tucatinib, and Trastuzumab in Patients With Metastatic, HER2+ Breast Cancer and a Multicenter, Randomized, Open-Label, Phase 2 Study of Preoperative Treatment With Ribociclib,Ttrastuzumab, Tucatinib, and Fulvestrant Versus Docetaxel, Carboplatin,Ttrastuzumab, and Pertuzumab in HR+/HER2+ Breast Cancer and Ribociclib, Trastuzumab, and Tucatinib Versus Docetaxel, Carboplatin, Trastuzumab, and Pertuzumab in Patients With HR-/HER2+ Breast Cancer
Brief Title: Ribociclib, Tucatinib, and Trastuzumab for the Treatment of HER2 Positive Breast Cancer
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Jonsson Comprehensive Cancer Center (Other)
Collaborators: Seagen Inc. (Industry); Novartis (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 21-001819; NCI-2021-11707 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2022-03-18; First posted 2022-04-08 (Actual); Last update posted 2025-05-13 (Actual); Status verified 2025-05

CONDITIONS: Anatomic Stage II Breast Cancer AJCC v8; Anatomic Stage IIA Breast Cancer AJCC v8; Anatomic Stage IIB Breast Cancer AJCC v8; Anatomic Stage III Breast Cancer AJCC v8; Anatomic Stage IIIA Breast Cancer AJCC v8; Anatomic Stage IIIB Breast Cancer AJCC v8; Anatomic Stage IIIC Breast Cancer AJCC v8; Anatomic Stage IV Breast Cancer AJCC v8; Invasive Breast Carcinoma; Locally Advanced HER2-Positive Breast Carcinoma; Metastatic HER2-Positive Breast Carcinoma; Prognostic Stage IB Breast Cancer AJCC v8; Prognostic Stage II Breast Cancer AJCC v8; Prognostic Stage IIA Breast Cancer AJCC v8; Prognostic Stage IIB Breast Cancer AJCC v8; Prognostic Stage III Breast Cancer AJCC v8; Prognostic Stage IIIA Breast Cancer AJCC v8; Prognostic Stage IIIB Breast Cancer AJCC v8; Prognostic Stage IIIC Breast Cancer AJCC v8; Prognostic Stage IV Breast Cancer AJCC v8
MeSH Terms: interventions — Carboplatin; Docetaxel; Fulvestrant; pertuzumab; 2C4 antibody; ribociclib; Trastuzumab; PF-05280014; Ogivri; Ontruzant; trastuzumab biosimilar HLX02; tucatinib

STUDY DESIGN:
Intervention Model Description: Phase Ib: Sequential assignment to increasing doses of ribociclib with fixed doses of tucatinib and trastuzumab.
  Phase II: Randomized assignment to 3 parallel arms.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (4):
- Phase Ib (ribociclib, tucatinib, trastuzumab) (Experimental): Patients receive ribociclib PO QD on days 1-21, tucatinib PO BID on days 1-28, and trastuzumab IV over 30-90 minutes every 7 days. Cycles repeat every 28 days for up to 4 cycles in the absence of disease progression or unacceptable toxicity.
  Interventions: Other: Quality-of-Life Assessment; Drug: Ribociclib; Biological: Trastuzumab; Drug: Tucatinib
- Phase II, Arm C (ribociclib, tucatinib, trastuzumab) (Experimental): Patients receive ribociclib PO QD on days 1-21, tucatinib BID on days 1-28, and trastuzumab IV over 30-90 minutes every 7 days. Cycles repeat every 28 days for up to 6 cycles in the absence of disease progression or unacceptable toxicity.
  Interventions: Other: Quality-of-Life Assessment; Drug: Ribociclib; Biological: Trastuzumab; Drug: Tucatinib
- Phase II,Arm A(ribociclib,tucatinib, trastuzumab, fulvestrant) (Experimental): Patients receive ribociclib PO QD on days 1-21, tucatinib BID on days 1-28, trastuzumab IV over 30-90 minutes every 7 days and fulvestrant subcutaneously (SC) on days 1 and 15 of cycle 1 and day 1 of every subsequent cycle. Cycles repeat every 28 days for up to 6 cycles in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Fulvestrant; Drug: Ribociclib; Biological: Trastuzumab; Drug: Tucatinib
- Phase II,Arm B(docetaxel,carboplatin,trastuzumab,pertuzumab) (Active Comparator): Patients receive docetaxel IV over 1 hour on day 1, carboplatin IV on day 1, trastuzumab IV over 30-90 minutes on day 1, and pertuzumab IV over 1 hour on day 1. Cycles repeat every 21 days for up to 6 cycles in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Carboplatin; Drug: Docetaxel; Biological: Pertuzumab; Other: Quality-of-Life Assessment; Biological: Trastuzumab

INTERVENTIONS:
Drug: Carboplatin — Given IV
  Other Names: Blastocarb; Carboplat; Carboplatin Hexal; Carboplatino; Carboplatinum; Carbosin; Carbosol; Carbotec; CBDCA; Displata; Ercar; JM-8; Nealorin; Novoplatinum; Paraplatin; Paraplatin AQ; Paraplatine; Platinwas; Ribocarbo
  Arms: Phase II,Arm B(docetaxel,carboplatin,trastuzumab,pertuzumab)
Drug: Docetaxel — Given IV
  Other Names: Docecad; RP56976; Taxotere; Taxotere Injection Concentrate
  Arms: Phase II,Arm B(docetaxel,carboplatin,trastuzumab,pertuzumab)
Drug: Fulvestrant — Given SC
  Other Names: Faslodex; Faslodex(ICI 182,780); ICI 182,780; ICI 182780; ZD9238
  Arms: Phase II,Arm A(ribociclib,tucatinib, trastuzumab, fulvestrant)
Biological: Pertuzumab — Given IV
  Other Names: 2C4; 2C4 Antibody; HS627; MoAb 2C4; Monoclonal Antibody 2C4; Omnitarg; Perjeta; Pertuzumab Biosimilar HS627; rhuMAb2C4; RO4368451
  Arms: Phase II,Arm B(docetaxel,carboplatin,trastuzumab,pertuzumab)
Other: Quality-of-Life Assessment — Ancillary Studies
  Other Names: Quality of Life Assessment
  Arms: Phase II, Arm C (ribociclib, tucatinib, trastuzumab); Phase II,Arm B(docetaxel,carboplatin,trastuzumab,pertuzumab); Phase Ib (ribociclib, tucatinib, trastuzumab)
Drug: Ribociclib — Given PO
  Other Names: Kisqali; LEE-011; LEE011
  Arms: Phase II, Arm C (ribociclib, tucatinib, trastuzumab); Phase II,Arm A(ribociclib,tucatinib, trastuzumab, fulvestrant); Phase Ib (ribociclib, tucatinib, trastuzumab)
Biological: Trastuzumab — Given IV
  Other Names: ABP 980; ALT02; Anti-c-ERB-2; Anti-c-erbB2 Monoclonal Antibody; Anti-ERB-2; Anti-erbB-2; Anti-erbB2 Monoclonal Antibody; Anti-HER2/c-erbB2 Monoclonal Antibody; Anti-p185-HER2; c-erb-2 Monoclonal Antibody; HER2 Monoclonal Antibody; Herceptin; Herceptin Biosimilar PF-05280014; Herceptin Trastuzumab Biosimilar PF-05280014; Herzuma; Kanjinti; MoAb HER2; Monoclonal Antibody c-erb-2; Monoclonal Antibody HER2; Ogivri; Ontruzant; PF-05280014; rhuMAb HER2; RO0452317; SB3; Trastuzumab Biosimilar ABP 980; Trastuzumab Biosimilar ALT02; trastuzumab biosimilar EG12014; Trastuzumab Biosimilar HLX02; Trastuzumab Biosimilar PF-05280014; Trastuzumab Biosimilar SB3; Trastuzumab Biosimilar SIBP-01; Trastuzumab-anns; Trastuzumab-dkst; Trastuzumab-dttb; Trastuzumab-pkrb; Trastuzumab-qyyp; Trazimera
Drug: Tucatinib — Given PO
  Other Names: ARRY-380; Irbinitinib; ONT-380; Tukysa
  Arms: Phase II, Arm C (ribociclib, tucatinib, trastuzumab); Phase II,Arm A(ribociclib,tucatinib, trastuzumab, fulvestrant); Phase Ib (ribociclib, tucatinib, trastuzumab)

SUMMARY:
This phase Ib/II trial studies the side effects and best dose of ribociclib, tucatinib, and trastuzumab for the treatment of HER2 positive breast cancer that has spread to other parts of the body (metastatic), and then compares the effect of ribociclib, tucatinib, trastuzumab with or without fulvestrant to docetaxel, carboplatin, trastuzumab, and pertuzumab (standard of care) for the treatment of early stage breast cancer before surgery (neoadjuvant therapy). Ribociclib and tucatinib may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Trastuzumab is a form of targeted therapy because it attaches itself to specific molecules (receptors) on the surface of tumor cells, known as HER2 receptors. When trastuzumab attaches to HER2 receptors, the signals that tell the cells to grow are blocked and the tumor cell may be marked for destruction by the body's immune system. Pertuzumab is a monoclonal antibody that may interfere with the ability of tumor cells to grow and spread. Estrogen can cause the growth of breast tumor cells. Fulvestrant blocks the use of estrogen by the tumor cells. Chemotherapy drugs, such as docetaxel and carboplatin, work in different ways to stop the growth of tumor cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Giving ribociclib, tucatinib, and trastuzumab with or without fulvestrant before surgery may make the tumor smaller and may reduce the amount of normal tissue that needs to be removed.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To assess the safety of the combination of ribociclib, tucatinib, and trastuzumab in patients with metastatic, HER2+ breast cancer. (Phase 1 Dose Escalation Trial) II. To determine the recommended phase 2 dose of ribociclib when combined with tucatinib and trastuzumab. (Phase 1 Dose Escalation Trial) III. To assess the pathologic complete response (pCR). (Phase 2 Neoadjuvant Study)

SECONDARY OBJECTIVES:

I. To evaluate the pharmacokinetics of ribociclib and tucatinib when given in combination. (Phase 1 Dose Escalation Trial) II. To assess the clinical objective response rate after 3 cycles via Response Evaluation Criteria in Solid Tumors (RECIST) 1.1. (Phase 1 Dose Escalation Trial) III. To assess the clinical objective response rate in the experimental arms. (Phase 2 Neoadjuvant Study) IV. To assess quality of life by evaluating toxicity burden using a quality of life (QOL)/patient-reported outcomes (PRO) questionnaire- the European Organization for Research and Treatment of Cancer Quality-of-Life Questionnaire-Core 30 (EORTC QLQ-C30) instrument. (Phase 2 Neoadjuvant Study) V. To assess the molecular changes in tumor biomarkers after 1 cycle of targeted therapy (anti-HER2, anti-estrogen, and CDK 4/6 directed therapy). (Phase 2 Neoadjuvant Study) VI. Pathological Assessment According to Residual Cancer Burden (RCB) Index at surgery. (Phase 2 Neoadjuvant Study)

EXPLORATORY OBJECTIVE:

I. To investigate potential serum and tumor predictive biomarkers to predict response to experimental therapy. (Phase 2 Neoadjuvant Study)

OUTLINE: This is a phase Ib, dose-escalation study of ribociclib followed by a phase II study.

PHASE Ib: Patients receive ribociclib orally (PO) once daily (QD) on days 1-21, tucatinib PO twice daily (BID) on days 1-28, and trastuzumab intravenously (IV) over 30-90 minutes every 7 days. Cycles repeat every 28 days for up to 4 cycles in the absence of disease progression or unacceptable toxicity.

PHASE II: Patients with hormone receptor (HR) positive status are randomized to Arm A or Arm B. Patients with HR negative status are randomized to Arm B or Arm C.

ARM A: Patients receive ribociclib PO QD on days 1-21, tucatinib BID on days 1-28, trastuzumab IV over 30-90 minutes every 7 days and fulvestrant subcutaneously (SC) on days 1 and 15 of cycle 1 and day 1 of every subsequent cycle. Cycles repeat every 28 days for up to 6 cycles in the absence of disease progression or unacceptable toxicity.

ARM B: Patients receive docetaxel IV over 1 hour on day 1, carboplatin IV on day 1, trastuzumab IV over 30-90 minutes on day 1, and pertuzumab IV over 1 hour on day 1. Cycles repeat every 21 days for up to 6 cycles in the absence of disease progression or unacceptable toxicity.

ARM C: Patients receive ribociclib PO QD on days 1-21, tucatinib BID on days 1-28, and trastuzumab IV over 30-90 minutes every 7 days. Cycles repeat every 28 days for up to 6 cycles in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed-up within 7 and 30 days.

ELIGIBILITY:
Inclusion Criteria:

* PHASE IB AND II: Patients over age of 18
* PHASE IB AND II: Available archival tissue for confirmatory central HER2 testing. Results not required prior to enrollment.
* PHASE IB AND II: Left ventricular ejection fraction (LVEF) >= 50% based on echocardiogram or multigated acquisition (MUGA).
* PHASE IB AND II: Platelet count >= 100,000/mm^3 (within 7 days before enrollment)

  * For Phase Ib only: Phase Ib allows for red blood cell transfusion, filgrastim (G-CSF), and hydration to meet eligibility requirements at the discretion of the investigator
* PHASE IB AND II: Hemoglobin >= 9.0 g/dL (within 7 days before enrollment)

  * For Phase Ib only: Phase Ib allows for red blood cell transfusion, G-CSF, and hydration to meet eligibility requirements at the discretion of the investigator
* PHASE IB AND II: Absolute neutrophil count (ANC) >= 1500/mm^3 (within 7 days before enrollment)

  * For Phase Ib only: Phase Ib allows for red blood cell transfusion, G-CSF, and hydration to meet eligibility requirements at the discretion of the investigator
* PHASE IB AND II: Creatinine clearance >= 30 mL/min as calculated using the Cockcroft-Gault equation or Serum creatinine =< 1.5 × upper limit of normal (ULN) (within 7 days before enrollment)

  * For Phase Ib only: Phase Ib allows for red blood cell transfusion, G-CSF, and hydration to meet eligibility requirements at the discretion of the investigator
* PHASE IB AND II: Alanine aminotransferase (ALT) < 2.5 × ULN, except for patients with liver metastasis, who are only included if the ALT is < 5 × ULN (within 7 days before enrollment)
* PHASE IB AND II: Aspartate aminotransferase (AST) < 2.5 × ULN, except for patients with liver metastasis, who are only included if the AST is < 5 × ULN (within 7 days before enrollment)
* PHASE IB AND II: Total bilirubin =< 1.5 x ULN. Participants with Gilbert's syndrome with a total bilirubin =< 2.0 times ULN and direct bilirubin within normal limits are permitted (within 7 days before enrollment)
* PHASE IB AND II: Serum Albumin >= 2.5 g/dL (within 7 days before enrollment)
* PHASE IB AND II: International normalized ratio (INR)/prothrombin time (PT) and activated partial thromboplastin time (aPTT) =< 1.5 × ULN (within 7 days before enrollment)
* PHASE IB AND II: Potassium within normal limits or corrected to within normal limits prior to first dose
* PHASE IB AND II: Magnesium within normal limits or corrected to within normal limits prior to first dose
* PHASE IB AND II: Total calcium (corrected for serum albumin) within normal limits or corrected to within normal limits prior to first dose
* PHASE IB AND II: Willingness and ability to comply with scheduled visits, treatment plans, laboratory tests, and other study procedures
* PHASE IB AND II: Patient can be premenopausal, perimenopausal, or post-menopausal at the time of study entry.

  * Premenopausal status is defined as either:

    * Patient had last menstrual period within the last 12 months, OR
    * If on tamoxifen or toremifene, plasma estradiol and follicle stimulating hormone (FSH) are in the premenopausal ranges according to central/local laboratory definition, OR
    * In case of therapy-induced amenorrhea, plasma estradiol and/or FSH are in the premenopausal ranges according to central/local laboratory definition

      * Perimenopausal status is defined as neither premenopausal nor postmenopausal
      * Postmenopausal is defined as not meeting premenopausal status
      * For pre-menopausal patients: Confirmed negative serum pregnancy test (beta-hCG) before starting study treatment or patient has had a hysterectomy. Male and female participants of reproductive/childbearing potential must agree to use a highly effective form of contraception or avoid intercourse during and upon completion of the study and for at least 7 months for females and 4 months for males after the last dose of study drug
* PHASE IB AND II: Male and female participants of reproductive/childbearing potential must agree to use a highly effective form of contraception or avoid intercourse during and upon completion of the study and for at least 7 months for females and 4 months for males after the last dose of study drug. Highly effective contraception methods include:

  * Total abstinence (when this is in line with the preferred and usual lifestyle of the patient). Periodic abstinence (e.g. calendar, ovulation, symptothermal, post-ovulation methods) and withdrawal are not acceptable methods of contraception
  * Double barrier method of contraception. The following are considered adequate barrier methods of contraception, must use 2: diaphragm, condom (by the partner), sponge, or spermicide/spermicidal jelly.
  * Female sterilization (have had surgical bilateral oophorectomy with or without hysterectomy), total hysterectomy or tubal ligation at least 6 weeks before taking trial treatment. In case of oophorectomy alone, only when the reproductive status of the woman has been confirmed by follow up hormone level assessment.
  * Male partner sterilization (at least 6 months prior to randomization). For female patients on the trial the vasectomized male partner should be the sole partner for that patient. If vasectomy of the male partner is the highly effective method of contraception chosen, the success of the vasectomy should be medically confirmed according to local practice
  * Placement of an intrauterine device (IUD)
* PHASE IB: Locally advanced/non-operable or metastatic HER2/neu amplified breast cancer, defined as 3+ by immunohistochemistry (IHC), or IHC 2+ and fluorescence in situ hybridization (FISH) + breast cancer
* PHASE IB: Received 1 or more prior lines of HER2 directed therapy in the metastatic setting
* PHASE IB: Recommended by the patient's treating oncologist to receive a tucatinib containing regimen as part of the next standard of care (SOC) line of therapy
* PHASE IB: Eastern Cooperative Oncology Group (ECOG) performance status 0-2
* PHASE IB: Measurable or non-measurable disease per RECIST 1.1
* PHASE IB: Based on screening contrast brain magnetic resonance imaging (MRI), patients must have one of the following:

  * No evidence of brain metastases
  * Untreated brain metastases not needing immediate local therapy. For patients with untreated central nervous system (CNS) lesions > 2.0 cm on screening contrast brain MRI, discussion with and approval from the medical monitor is required prior to enrollment
  * Previously treated brain metastases

    * Brain metastases previously treated with local therapy may either be stable since treatment or may have progressed since prior local CNS therapy, provided that there is no clinical indication for immediate re-treatment with local therapy in the opinion of the investigator
    * Patients treated with CNS local therapy for newly identified lesions found on contrast brain MRI performed during screening for this study may be eligible to enroll if all of the following criteria are met:

      * Time since whole-brain radiotherapy (WBRT) is >= 21 days prior to first dose of treatment, time since stereotactic radiosurgery (SRS) is >= 7 days prior to first dose of treatment, or time since surgical resection is >= 28 days
      * Other sites of disease assessable by RECIST 1.1 are present
  * Relevant records of any CNS treatment must be available to allow for classification of target and non-target lesions
* PHASE II: Operable HER2/neu amplified invasive breast cancer, defined as 3+ by IHC, or IHC 2+ and FISH +
* PHASE II: Known Ki67 status
* PHASE II: Previously untreated operable invasive carcinoma of the breast greater than 2.0 cm (cT2) in size based on imaging or physical exam or imaging. Patients with clinical node negative disease or clinical node (cN1/cN2) positive are allowed provided they are deemed to have operable disease at study entry
* PHASE II: Patients with clinically involved lymph nodes should not have evidence of distant disease based on standard of care staging imaging prior to informed consent form (ICF) signature
* PHASE II: Breast cancer suitable for mandatory baseline core biopsy
* PHASE II: No prior systemic therapy or radiotherapy for currently-diagnosed invasive or non-invasive breast cancer
* PHASE II: Eastern Cooperative Oncology Group (ECOG) performance status 0-1

Exclusion Criteria:

* PHASE IB AND II: Concurrent therapy with any other non-protocol anti-cancer therapy
* PHASE IB AND II: History of any other malignancy within the past 5 years, with the exception of non-melanoma skin cancer or carcinoma-in-situ of the cervix
* PHASE IB AND II: Proteinuria estimated by urine protein: creatinine ratio > 3.5 on a random urine sample
* PHASE IB AND II: Uncontrolled arterial hypertension despite optimal medical management
* PHASE IB AND II: Patient has known active hepatitis B virus (HBV) or hepatitis C virus (HCV), or Human immunodeficiency virus (HIV) infection (testing is not mandatory, unless required by local regulation)
* PHASE IB AND II: Uncontrolled infection; active, clinically serious infections (> Common Terminology Criteria for Adverse Events [CTCAE] grade 2)
* PHASE IB AND II: Clinically significant, uncontrolled heart disease and/or cardiac repolarization abnormality, including any of the following:

  * History of documented myocardial infarction (MI), angina pectoris, symptomatic pericarditis, or coronary artery bypass graft (CABG) within 6 months prior to study entry
  * Documented cardiomyopathy
  * Left ventricular ejection fraction (LVEF) < 50% as determined by multiple gated acquisition (MUGA) scan or echocardiogram (ECHO)
  * Long QT syndrome or family history of idiopathic sudden death or congenital long QT syndrome, or any of the following:

    * Risk factors for Torsades de Pointe (TdP) including uncorrected hypocalcemia, hypokalemia or hypomagnesemia, history of cardiac failure, or history of clinically significant/symptomatic bradycardia
    * Concomitant medication(s) with a known risk to prolong the QT interval and/or known to cause Torsades de Pointe that cannot be discontinued or replaced by safe alternative medication (e.g., within 5 half-lives or 7 days prior to starting study drug)
    * Inability to determine the corrected QT using Fridericia's formula (QTcF) interval
    * Clinically significant cardiac arrhythmias (e.g., ventricular tachycardia), complete left bundle branch block, high-grade atrioventricular (AV) block (e.g., bifascicular block, Mobitz type II and third degree AV block)
    * Systolic blood pressure (SBP) > 160 or < 90 mmHg
* PHASE IB AND II: Congestive heart failure > New York Heart Association (NYHA) class 2
* PHASE IB AND II: History of baseline QT prolongation > 450 msec
* PHASE IB AND II: Unstable angina (angina symptoms at rest), new-onset angina (begun within the last 3 months)
* PHASE IB AND II: Myocardial infarction less than 6 months before start of test drug
* PHASE IB AND II: Anti-arrhythmic therapy (beta blockers or digoxin are permitted)
* PHASE IB AND II: Arterial or venous thrombotic or embolic events such as cerebrovascular accident (including transient ischemic attacks), deep vein thrombosis or pulmonary embolism within 3 months before the start of study medication.
* PHASE IB AND II: Participants receiving anticoagulation therapy are not allowed
* PHASE IB AND II: Patients with evidence or history of bleeding diathesis. Any hemorrhage or bleeding event >= CTCAE Grade 3 within 4 weeks of start of study medication
* PHASE IB AND II: Non-healing wound or ulcer
* PHASE IB AND II: History of, or current autoimmune disease (other than Hashimoto's thyroiditis with normal thyroid stimulating hormone [TSH])
* PHASE IB AND II: Major surgical procedure or significant traumatic injury (as judged by the investigator) within 28 days before start of study medication, open biopsy within 7 days before start of study medication
* PHASE IB AND II: Unable to swallow pills or has significant gastrointestinal disease which would preclude the adequate oral absorption of medications
* PHASE IB AND II: Patients with seizure disorder requiring medication
* PHASE IB AND II: Known hypersensitivity to any of the study drugs, study drug classes, or excipients in the formulation
* PHASE IB AND II: Systemic continuous corticosteroid therapy at a daily dose higher than 15 mg prednisone or equivalent is not allowed. Patients may be using topical or inhaled corticosteroids. Previous corticosteroid therapy must be stopped or reduced to the allowed dose at least 7 days prior to the first study drug administration. If a patient is on chronic corticosteroid therapy, corticosteroids should be de-escalated to the maximum allowed dose after the patient has signed the consent document
* PHASE IB AND II: History of having received an allogeneic bone marrow or organ transplant
* PHASE IB AND II: Chronic oxygen therapy
* PHASE IB AND II: Use of a strong cytochrome P450 (CYP)2C8 inhibitor within 5 half-lives of the inhibitor or use of a strong CYP3A4 or CYP2C8 inducer within 5 days prior to the first dose of study treatment
* PHASE IB: Early stage (curable) breast cancer
* PHASE IB: Based on screening brain MRI, patients must not have any of the following:

  * Any untreated brain lesions > 2.0 cm in size, unless discussed with medical monitor and approval for enrollment is given
  * Ongoing use of systemic corticosteroids for control of symptoms of brain metastases at a total daily dose of > 2 mg of dexamethasone (or equivalent). However, patients on a chronic stable dose of =< 2 mg total daily of dexamethasone (or equivalent) may be eligible with discussion and approval by the medical monitor
  * Any brain lesion thought to require immediate local therapy, including (but not limited to) a lesion in an anatomic site where increase in size or possible treatment-related edema may pose risk to patient (e.g. brain stem lesions). Patients who undergo local treatment for such lesions identified by screening contrast brain MRI may still be eligible for the study based on criteria described under CNS inclusion criteria
* PHASE IB: Known or suspected leptomeningeal disease (LMD) as documented by the investigator
* PHASE IN: Have poorly controlled (> 1/week) generalized or complex partial seizures, or manifest neurologic progression due to brain metastases notwithstanding CNS-directed therapy
* PHASE II: Metastatic breast cancer (local spread to axillary or internal mammary lymph nodes is permitted)
* PHASE II: Current therapy with raloxifene, tamoxifen, aromatase inhibitor, or other selective estrogen receptor modulator (SERM), gonadotrophin-releasing hormone (GNRH) agonist/antagonist, either for osteoporosis or prevention of breast cancer. Subjects must have discontinued therapies for at least 28 days prior to first baseline biopsy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2022-04-07 (Actual); Primary Completion 2026-04-01 (Estimated); Study Completion 2027-04-01 (Estimated)

PRIMARY OUTCOMES:
Maximum tolerated dose (MTD) (Phase Ib) | During the first cycle of treatment (1 cycle = 28 days)
  Defined as the highest dose level that does not lead to unacceptable toxicity in two or more patients in a dosing level.
Pathologic complete response (pCR) (Phase II) | Up to 30 days after last treatment dose
  Defined as no invasive tumor in the breast or lymph nodes at the time of surgery. Response evaluable participants are defined as participants who are randomized and have receive at least one cycle of protocol therapy. The pCR rate is defined as percentage of randomized patients with a pCR in each of the treatment arms.The estimated pCR rate (and 95% confidence interval [CIs]) will be calculated for each experimental arm and compared to the corresponding control arm using the Cochran-Mantel-Haenszel x^2 test, with a two-sided significance level of 5%. Absolute differences in pCR rate between study arms will be calculated, along with 95% exact confidence intervals. This will be stratified according to hormone receptor (HR) status Multivariate logistic regression will be used to control for important baseline characteristics and odds ratios with corresponding CIs will be calculated.

SECONDARY OUTCOMES:
Clinical objective response rate (ORR) (Phase IB and II) | Up to 30 days after last treatment dose
  ORR will be evaluated by Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 using caliper measurements. A responder is defined as any participant who exhibits a complete response (CR) or partial response (PR). The clinical response rate is estimated as the total number of CRs and PRs divided by the total number of participants randomized.The estimated ORR rate (and 95% CIs) will be calculated for each treatment arm and compared using the Cochran-Mantel-Haenszel x^2 test, with a two-sided significance level of 5%. Absolute differences in pCR rate between study arms will be calculated, along with 95% exact confidence intervals. This will be stratified according to HR status. Multivariate logistic regression will be used to control for important baseline characteristics and odds ratios with corresponding CIs will be calculated.
Evaluate the pharmacokinetics of ribociclib and tucatinib when given in combination with tucatinib and trastuzumab. (Phase 1b): Area Under Curve (AUC) | Pre-infusion and 1, 2, 3, and 6 hours after the start of the infusion
  The pharmacokinetic (PK) parameter - area under the plasma concentration-time curve (AUC) will be determined for ribociclib and tucatinib in all Phase 1b participants.
Evaluate the pharmacokinetics of ribociclib and tucatinib when given in combination with tucatinib and trastuzumab. (Phase 1b): Elimination half-life (t½) | Pre-infusion and 1, 2, 3, and 6 hours after the start of the infusion
  The pharmacokinetic (PK) parameter - Elimination half-life (t½) will be determined for for ribociclib and tucatinib in all Phase 1b participants.
Evaluate the pharmacokinetics of ribociclib and tucatinib when given in combination with tucatinib and trastuzumab. (Phase 1b): Maximum plasma concentration (Cmax) | Pre-infusion and 1, 2, 3, and 6 hours after the start of the infusion
  Maximum plasma concentration (Cmax) will be determined for for ribociclib and tucatinib in all Phase 1b participants.
Evaluate the pharmacokinetics of ribociclib and tucatinib when given in combination with tucatinib and trastuzumab. (Phase 1b): Minimum plasma concentration | Pre-infusion and 1, 2, 3, and 6 hours after the start of the infusion
  Minimum plasma concentration will be determined for ribociclib and tucatinib in all Phase 1b participants.
Evaluate the pharmacokinetics of ribociclib and tucatinib when given in combination with tucatinib and trastuzumab. (Phase 1b): Time when Cmax occurs (Tmax) | Pre-infusion and 1, 2, 3, and 6 hours after the start of the infusion
  Time when Cmax occurs (Tmax) will be determined for ribociclib and tucatinib in all Phase 1b participants.
Evaluate the pharmacokinetics of ribociclib and tucatinib when given in combination with tucatinib and trastuzumab. (Phase 1b): Average plasma concentration at steady state (Cavg) | Pre-infusion and 1, 2, 3, and 6 hours after the start of the infusion
  Average plasma concentration at steady state (Cavg) will be determined for ribociclib and tucatinib in all Phase 1b participants.
Quality of life (QOL) (Phase II) | Up to 7 days after last treatment dose
  The EPRTC QLQ-C30 (European Organization for the Research and Treatment of Cancer- Quality of Life questionnaire) is composed of both multi-item scales and single-item measures. These include five functional scales, three symptom scales, a global health status / Quality of Life (QoL) scale, and six single items. Each of the multi-item scales includes a different set of items - no item occurs in more than one scale.
  All of the scales and single-item measures range in score from 0 to 100. A high scale score represents a higher response level. Thus a high score for a functional scale represents a high / healthy level of functioning, a high score for the global health status / QoL represents a high QoL, but a high score for a symptom scale / item represents a high level of symptomatology / problems.
Measure the gene expression and/or biomarker changes that may be correlated with or predict biological, clinical, and pathologic response (Phase II) | Up to 30 days after last treatment dose
  Primary analysis of these molecular changes will include a linear model with treatment and hormone receptor status fixed effects. Separate analyses for change after 1 cycle and all cycles will be performed and compared to baseline levels. Serum and tumor biomarker analyses, including but not limited to on treatment tumor CD45 expression and germline IL6 promoter genotyping will be correlated with clinical outcomes and important clinical characteristics. Absolute change in Ki67 and cell cycle arrest rate (defined as a Ki67 of =< 2.7%) will be analyzed separately.

CONTACTS AND LOCATIONS:
Overall Officials: Nicholas P McAndrew, Principal Investigator — UCLA / Jonsson Comprehensive Cancer Center
Locations (1):
- UCLA / Jonsson Comprehensive Cancer Center, Los Angeles, California, United States